CLINICAL TRIAL: NCT05129371
Title: The Effect of Breathing Exercise on Fatigue in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Selva Ezgi Askar, Lecturer, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HMKUASKAR-01
Record Dates: First submitted 2021-10-25; First posted 2021-11-22 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure; Fatigue
Keywords: Fatigue; Heart Failure; Breathing exercise; Nursing
MeSH Terms: conditions — Heart Failure; Fatigue | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Patients willing to participate in the study are evaluated according to the inclusion and exclusion criteria. Afterwards, they are divided into 3 groups with the stratified sampling method. The intervention group is given face-to-face breathing exercises under the supervision of the trainer, through video calls over the WhatsApp application after discharge. The placebo group is asked to breathe normally through the nose with eyes closed, sitting in the same position as the intervention group, under the supervision of the trainer. Venous oxygen saturation, heart rate/minute and respiratory rate/minute are monitored by pulse oximetry given to the participants in the intervention and placebo groups before and after each session for 8 weeks. The severity of fatigue of the participants in all groups; It is measured before starting the application, in the middle of the application period (4th week) and after the application is completed (8th week).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breathing Exercise Group (Active Comparator): This group will be given breathing exercises in accordance with the determined protocol.
  Interventions: Other: Breathing exercise
- Placebo Breathing Group (Placebo Comparator): Normal breathing of this group will be monitored.
  Interventions: Other: Placebo Breathing Group
- Control Group (No Intervention): No application will be made to this group.

INTERVENTIONS:
Other: Breathing exercise — Following the protocol prepared, the breathing exercise group is given breathing exercises for about 20 minutes, 3 times a week for 8 weeks, under the supervision of the trainer, in the hospital face-to-face, and after discharge through video calls over the WhatsApp application. Reminders (by text message or voice call) are used for the remaining 4 days of the week, allowing the patient to do it on their own.
  Arms: Breathing Exercise Group
Other: Placebo Breathing Group — The placebo group is asked to breathe normally through the nose with eyes closed, sitting in the same position as the intervention group for 10-15 minutes, 3 times a week for 8 weeks, under the supervision of the trainer, in the hospital face-to-face, and after discharge through video calls over the WhatsApp application.
  Arms: Placebo Breathing Group

SUMMARY:
In this study, It is aimed to evaluate the effect of breathing exercise on fatigue in patients with heart failure, to reduce the severity of fatigue in participants, and thus to enable patients to participate more actively in daily life.

DETAILED DESCRIPTION:
In the Heart Failure Prevalence and Indicators study in Turkey, the prevalence of heart failure (HF) in the adult population was determined as 3.2%. In line with this study, although Turkey has a young population, it is seen that the prevalence of HF is higher than in western countries. As it is known, fatigue is one of the most characteristic symptoms of HF and it was determined that the perceived fatigue was moderate or severe in 92% of the patients. There is a decrease in the activities of daily living of patients with fatigue and their quality of life is adversely affected. For this reason, nurses have an active role in the evaluation of fatigue and in ensuring that the patient can cope with fatigue with appropriate interventions. In the management of fatigue, non-pharmacological approaches are frequently used in addition to current pharmacological treatment. Breathing exercises, one of the non-pharmacological approaches used; consists of breathing control and exercises that create body awareness. It also controls the instincts and the mind. In a study conducted with patients with multiple sclerosis; Upper extremity exercise and breathing exercises were combined as a home-based program, 2 days a week in 60-minute sessions. It has been demonstrated that the 4-week program contributes to the reduction of fatigue. However; A study reported to be the first to evaluate the effects of yoga and specific breathing techniques for improving cardiovascular function, autonomic system, and quality of life in heart failure patients with preserved ejection fraction is still in the patient selection and intervention stages. In this study, the participants were randomly divided into three groups, and active breathing techniques were applied to the first group and passive breathing techniques to the second group. The third group (control) receives standard pharmacological treatment. The application period is done in 45-minute sessions twice a week for 8 weeks. There is no study in the literature investigating the effect of breathing exercise on fatigue in patients with heart failure. In this study, which was planned in the light of this information; It is aimed to evaluate the effect of breathing exercise on fatigue in patients with heart failure, to reduce the severity of fatigue in patients, and thus to enable patients to participate more actively in daily life.

ELIGIBILITY:
Inclusion Criteria:

* Citizen of T.C.
* 18 years old and over
* Diagnosed with heart failure at least 6 months ago, according to the heart failure classification of the New York Heart Association (NYHA) II. or III. in phase
* Left ventricular ejection fraction < 50%
* Volunteer to participate in the research
* Piper fatigue scale score of 4 and above
* Hb value of 8 gm/dL or more
* Having an Internet connection and a smartphone at or near Patients meeting all of the above criteria are included in the study.

Exclusion Criteria:

* Those who are taking or doing yoga/pranayama/deep breathing exercises before diagnosis
* Having a problem (due to deviation of the septum, etc.) that causes difficulty in doing breathing exercises
* Have a serious mental illness/cognitive problem that may affect their perception or communication
* Receiving chemotherapy treatment
* Have had cardiovascular surgery in the last 3 months
* Those who have had myocardial infarction in the last 3 months
* Have had valve surgery in the last 6 months
* Have chronic obstructive pulmonary disease or asthma
* Chronic renal failure with glomerular filtration rate < 30 ml/min
* Have a serious disease related to heart valves
* Piper fatigue scale score below 4
* Hb value below 8 gm/dL
* Existing Cardiac Resynchronization Therapy (CRT)
* Implantable Cardioverter Defibrillator (ICD) administered in the past 6 months
* Those who were informed about the research but did not want to participate in the research

In case of any of the above criteria, the patient is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in fatigue | 2 months
  Fatigue severity is expected to change in the intervention group compared to the other groups. Fatigue severity will be measured with Piper Fatigue Scale at the end of the 1st and 2nd months. The Piper Fatigue Scale consists of 22 items, each of which is evaluated over time on a 0-10 point VAS (Visual Analog Scale), and evaluates the patient's subjective perception of fatigue with four sub-dimensions. Total fatigue score is obtained by summing the items and dividing by the total number of items. As a result of the average score, 0 points indicate no fatigue, 1-3 points indicate mild fatigue, 4-6 points indicate moderate fatigue, and 7-10 points indicate severe fatigue. It was determined that the items in the subgroup and the general scale were in a strong relationship, and the reliability coefficient was quite high, 0.94 in the general scale. As a result, it has been determined that this scale is reliable in evaluating the multidimensional perception of fatigue.

SECONDARY OUTCOMES:
Change in venous oxygen saturation | Up to 8 weeks
  Change in venous oxygen saturation is expected in the intervention group compared to the other groups. Venous oxygen saturation value will be measured before and after each session for 8 weeks.
Change in heart rate/minute | Up to 8 weeks
  Change in heart rate/minute is expected in the intervention group compared to the other groups. Heart rate/minute value will be measured before and after each session for 8 weeks.
Change in respiratory rate/minute | Up to 8 weeks
  Change in respiratory rate/minute is expected in the intervention group compared to the other groups. Respiratory rate/minute value will be measured before and after each session for 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Selva Ezgi Aşkar, Principal Investigator — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University Hospital, Hatay, Turkey (Türkiye)

REFERENCES:
- [Background] Degertekin M, Erol C, Ergene O, Tokgozoglu L, Aksoy M, Erol MK, Eren M, Sahin M, Eroglu E, Mutlu B, Kozan O. [Heart failure prevalence and predictors in Turkey: HAPPY study]. Turk Kardiyol Dern Ars. 2012 Jun;40(4):298-308. doi: 10.5543/tkda.2012.65031. Turkish. PMID 22951845
- [Background] Efe F., Olgun N. The Effect of Education on Dyspnea, Fatigue and Quality of Life in Patients with Heart Failure. Hacettepe University Faculty of Health Sciences Nursing Journal 2011; 1-13.
- [Background] Ovayolu O. Ovayolu N. Evidence in Yoga Practices. HUHEMFAD-JOHUFON 2019; 6 (1): 44-49.
- [Background] Grubic Kezele T, Babic M, Stimac D. Exploring the feasibility of a mild and short 4-week combined upper limb and breathing exercise program as a possible home base program to decrease fatigue and improve quality of life in ambulatory and non-ambulatory multiple sclerosis individuals. Neurol Sci. 2019 Apr;40(4):733-743. doi: 10.1007/s10072-019-3707-0. Epub 2019 Jan 18. PMID 30659416
- [Background] Lopes CP, Danzmann LC, Moraes RS, Vieira PJC, Meurer FF, Soares DS, Chiappa G, Guimaraes LSP, Leitao SAT, Ribeiro JP, Biolo A. Yoga and breathing technique training in patients with heart failure and preserved ejection fraction: study protocol for a randomized clinical trial. Trials. 2018 Jul 28;19(1):405. doi: 10.1186/s13063-018-2802-5. PMID 30055633